CLINICAL TRIAL: NCT06767579
Title: Comparison of the Incidence of Delirium Caused by Different Anesthetic Agents in Patients Undergoing Liver Transplantation
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-1084
Record Dates: First submitted 2024-11-28; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sevoflurane Inhalation Anesthesia Group: Sevoflurane Inhalation Anesthesia Group in Liver Transplantation Patients
- Propofol Intravenous Anesthesia Group: Propofol Intravenous Anesthesia Group in Liver Transplantation Patients

SUMMARY:
This study is a prospective observational study that analyzes the incidence of postoperative delirium in patients undergoing liver transplantation, based on the use of the inhalational anesthetic sevoflurane and the intravenous anesthetic propofol.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and older
* Patients undergoing liver transplantation who are scheduled to receive anesthesia with the inhaled anesthetic sevoflurane or the intravenous anesthetic propofol.

Exclusion Criteria:

* Individuals with hearing loss, cognitive impairment or obvious dementia, hepatic encephalopathy, or difficulty in communication.
* Diagnosed with neurological disorders (e.g., brain hemorrhage, stroke, dementia, Parkinson's disease, cognitive impairment, etc.).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adults aged 19 years or older
  * Recipients of liver transplants who are scheduled to undergo anesthesia using the inhalation anesthetic sevoflurane or the intravenous anesthetic propofol
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2028-10-17 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative delirium | from postoperative day 0 to postoperative day 7
  At least two times a day during the hospitalization period. Patients diagnosed with delirium using the CAM were evaluated for the duration, symptoms, and type of delirium (e.g., reduced awareness of the environment; poor cognitive skills; behavioral changes; and emotional disturbances).
  ** Confusion assessment methods(CAM) diagnostic algorism (positive or negative result, positive means delirium)
  CAM is considered positive if features 1 and 2 are present, with at least one of features 3 or 4. Below are the four criteria of features :
  1. Acute onset and fluctuating course Determined by collateral history or repeated clinic assessment
  2. Inattention Counting from 20-1 is a simple (if blunt) test for this
  3. Disorganized thinking
  4. Altered levels of consciousness

SECONDARY OUTCOMES:
comprehensive geriatric assessment(CGA) | Participants will be followed for the duration of their hospital stay and until their visit within one month after discharge, with an expected average of 4 weeks
  Core component of CGA are as follows :
  The Korean version of the fatigue, resistance, ambulation, illnesses, and loss of weight (K-FRAIL) scale : 0(healthy)~8(frail) Mini Nutritional Assessment(MNA) : 0 (malnutrition)~14(normal) Geriatric Depression Scale(GDS) : 0(normal)~ 15(depression) Instrumental Activities of Daily Living(IADL)-Lawton-Brody Scale : 0~8(complete independence)
duration of delirium | Participants will be followed for the duration of their hospital stay and until their visit within one month after discharge, with an expected average of 4 weeks
  Duration of Delirium: The duration of delirium is measured from the onset to the resolution of symptoms, recorded in hours or days (e.g., 1 day, 3 days, 5 days).
total score of QOR-40 | Participants will be followed for the duration of their hospital stay and until their visit within one month after discharge, with an expected average of 4 weeks
  The Quality of Recovery-40 (QoR-40) 40~200(better recovery)
type of delirium | Participants will be followed for the duration of their hospital stay and until their visit within one month after discharge, with an expected average of 4 weeks
  Type of Delirium: Delirium is classified into three types: hyperactive, hypoactive, and mixed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No